CLINICAL TRIAL: NCT00899626
Title: Novel Colon Cancer Markers in Gastrointestinal Tissue and Biofluids
Brief Title: Gastrointestinal Biomarkers in Tissue and Biological Fluid Samples from Colorectal Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kristen K Ciombor, Associate Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: CDR0000584214; P30CA068485 (NIH); VU-VICC-GI-0283 (Other: Vanderbilt University Medical Center); VU-VICC-010680 (Other: Vanderbilt University Medical Center)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer; Esophageal Cancer; Gastric Cancer; Pancreatic Cancer; Precancerous Condition
Keywords: colon cancer; gastric cancer; pancreatic cancer; esophageal cancer; adenomatous polyp
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Precancerous Conditions; Colonic Neoplasms; Adenomatous Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Tissue, Body Fluids
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
RATIONALE: Studying samples of tissue, blood, urine, stool, and other biological fluids from patients with cancer and from healthy volunteers undergoing colonoscopy or endoscopy may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This research study is looking at gastrointestinal biomarkers in tissue and biological fluid samples from patients and participants undergoing colonoscopy, endoscopy, or surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify new potential biomarkers of increased gastrointestinal cancer risk using tissue and biofluid samples from patients and volunteers undergoing colonoscopy, endoscopy, or surgery.
* Develop new screening strategies based on substances found in tissue and biofluid samples.

OUTLINE: This is a multicenter study.

Patients and healthy volunteers undergo colonoscopy, endoscopy, or surgery. Patients and healthy volunteers also undergo tissue (e.g., tumor or normal mucosa) and biofluid (e.g., blood, urine, cyst fluids or tumor cells, bile and pancreatic juices, and/or stool) sample collection. Samples are analyzed for tumor markers by proteomic methods and protein analysis. If candidate biomarkers are identified, samples are stored for future studies involving these biomarkers. Information, including demographics, personal and family history of cancer, and prior and current colonoscopy, endoscopy, or surgery results, is collected from the medical record and stored in the project database.

Patients are followed once a year for up to 5 years to determine if biomarkers have a prognostic significance.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing colonoscopy or endoscopy for diagnostic or screening purposes at the Vanderbilt University Medical Center or at the Veterans Affairs Medical Center AND
* Meets 1 of the following criteria:

  * Diagnosis of gastrointestinal (GI) cancer, polyps, or inflammatory bowel disease
  * History of previously treated GI cancer, polyps, or inflammatory bowel disease

PATIENT CHARACTERISTICS:

* Capable of giving informed consent
* Not mentally or medically impaired
* No bleeding disorder

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vanderbilt University Medical Center patients with GI malignancy
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2002-06; Primary Completion 2045-10 (Estimated); Study Completion 2045-10 (Estimated)

PRIMARY OUTCOMES:
Identification of new potential biomarkers of increased gastrointestinal cancer risk using tissue and biofluid samples from patients undergoing colonoscopy, endoscopy, or surgery | Through study completion, approximately 30 years
  Genomic and proteomic biomarkers
Development of new screening strategies based on substances found in tissue and biofluid samples | Through study completion, approximately 30 years
  Genomic and proteomic biomarker discovery

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Background] Smith JJ, Deane NG, Wu F, Merchant NB, Zhang B, Jiang A, Lu P, Johnson JC, Schmidt C, Bailey CE, Eschrich S, Kis C, Levy S, Washington MK, Heslin MJ, Coffey RJ, Yeatman TJ, Shyr Y, Beauchamp RD. Experimentally derived metastasis gene expression profile predicts recurrence and death in patients with colon cancer. Gastroenterology. 2010 Mar;138(3):958-68. doi: 10.1053/j.gastro.2009.11.005. Epub 2009 Nov 13. PMID 19914252
- [Background] Oh SC, Park YY, Park ES, Lim JY, Kim SM, Kim SB, Kim J, Kim SC, Chu IS, Smith JJ, Beauchamp RD, Yeatman TJ, Kopetz S, Lee JS. Prognostic gene expression signature associated with two molecularly distinct subtypes of colorectal cancer. Gut. 2012 Sep;61(9):1291-8. doi: 10.1136/gutjnl-2011-300812. Epub 2011 Oct 13. PMID 21997556
- [Background] Tripathi MK, Deane NG, Zhu J, An H, Mima S, Wang X, Padmanabhan S, Shi Z, Prodduturi N, Ciombor KK, Chen X, Washington MK, Zhang B, Beauchamp RD. Nuclear factor of activated T-cell activity is associated with metastatic capacity in colon cancer. Cancer Res. 2014 Dec 1;74(23):6947-57. doi: 10.1158/0008-5472.CAN-14-1592. Epub 2014 Oct 15. PMID 25320007
- [Background] Zhu J, Deane NG, Lewis KB, Padmanabhan C, Washington MK, Ciombor KK, Timmers C, Goldberg RM, Beauchamp RD, Chen X. Evaluation of frozen tissue-derived prognostic gene expression signatures in FFPE colorectal cancer samples. Sci Rep. 2016 Sep 14;6:33273. doi: 10.1038/srep33273. PMID 27623752